CLINICAL TRIAL: NCT01599585
Title: A Randomized Controlled Trial of In-Home Tele-behavioral Health Care Utilizing Behavioral Activation for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Telehealth and Technology (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-11-2-0118; W81XWH-11-2-0118 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity)
Record Dates: First submitted 2012-05-11; First posted 2012-05-16 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Depression
Keywords: Depression; Behavioral Activation; Tele-medicine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In Home (Experimental): Participants in this condition will receive 8 sessions of BA treatment over the course of approximately 8 weeks (one session per week). The sessions will be conducted in their homes using an Army approved secure web-based video conferencing system. BA has been successfully delivered in this time frame, and it has been delivered via in-home video conferencing technology.
  Interventions: Behavioral: Behavioral Activation
- In-Person (Active Comparator): Participants in this condition will receive 8 sessions of BA treatment over the course of approximately 8 weeks (one session per week with allowance for rescheduled sessions). The sessions will be conducted in a clinic setting at The National Center for Telehealth & Technology.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral activation(BA)will be delivered in 8 weekly sessions via webcam for the in-home arm or face to face in the in-person arm. Behavioral activation attempts to help depressed individuals reengage in their lives through focused activation strategies.
  Other Names: BA

SUMMARY:
This study will evaluate the effectiveness of a web-based behavioral activation(BA) treatment for depression by comparing it to in-person BA treatment in Soldiers and Veterans with Major and Minor Depressive Disorder. We will test the hypothesis that 8 sessions of in-home BA delivered via a webcam will be as safe and effective in reducing symptoms of hopelessness and depression as in-person BA treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

* Current Major Depressive or Minor Depressive Disorder
* High-speed internet/network access at home (384kbs minimum)
* Informed consent
* Fluent in the English language

Exclusion Criteria:

* Currently undergoing psychotherapy for depression
* less than 18 or greater than 65 year of age
* Active psychotic symptoms/disorders as determined by the SCID for DSM-IV
* Dysthymic Disorder
* Current suicidal ideation with intent or recent (within six months) history of a suicide attempt
* History of Organic Mental Disorder
* Current substance dependence as determined by the SCID (lifetime substance dependence or substance abuse will not be excluded)
* History of violence or poor impulse control causing potential risk to staff or others
* Significant ongoing stressors that require urgent crisis intervention
* Having a living arrangement that will not permit the use of a private space to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Gahm, PhD, Principal Investigator — National Center for Telehealth and Technology; David D Luxton, PhD, Principal Investigator — National Center for Telehealth & Technology
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, Oregon
  - National Center for Telehealth and Technology, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewinsohn PM, Graf M. Pleasant activities and depression. J Consult Clin Psychol. 1973 Oct;41(2):261-8. doi: 10.1037/h0035142. No abstract available. PMID 4147832
- [Background] Egede LE, Frueh CB, Richardson LK, Acierno R, Mauldin PD, Knapp RG, Lejuez C. Rationale and design: telepsychology service delivery for depressed elderly veterans. Trials. 2009 Apr 20;10:22. doi: 10.1186/1745-6215-10-22. PMID 19379517
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Freedland KE, Skala JA, Carney RM, Rubin EH, Lustman PJ, Davila-Roman VG, Steinmeyer BC, Hogue CW Jr. Treatment of depression after coronary artery bypass surgery: a randomized controlled trial. Arch Gen Psychiatry. 2009 Apr;66(4):387-96. doi: 10.1001/archgenpsychiatry.2009.7. PMID 19349308
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Mackenzie CS, Gekoski WL, Knox VJ. Age, gender, and the underutilization of mental health services: the influence of help-seeking attitudes. Aging Ment Health. 2006 Nov;10(6):574-82. doi: 10.1080/13607860600641200. PMID 17050086
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] King R. Cognitive therapy of depression. Aaon Beck, John Rush, Brian Shaw, Gary Emery. New York: Guilford, 1979. Aust N Z J Psychiatry. 2002 Apr;36(2):272-5. doi: 10.1046/j.1440-1614.2002.t01-4-01015.x. No abstract available. PMID 11982560
- [Background] Lewinsohn, PM, Biglan, A, Zeiss, AS. Behavioral treatment of depression. The behavioral management of anxiety, depression and pain. (pp.91-46. New York; Bunner/Mazel
- [Background] Lewinsohn, PM, Gotlib, IH. Behavioral theory and treatment of depression. In E.E. Beckham and W.R. Leber (Eds). Handbook of depression (pp.352-375) New York: Guildford, 1995
- [Background] Jacobson, NS, Martell, CR and Dimidjian, S. Behavioral activation therapy for depression: Returning to contextual roots. Clinical Psychology: Science and Practice 8(3):255-270, 2002
- [Background] First, MB, Spitzer RL, Gibbon, M and Williams, JBW. Structured Clinical Interview for DSM-IV Axis Disorders. Arlington, VA: American Psychiatric Press. 2002
- [Background] Hopko DR, Lejuez CW, LePage JP, Hopko SD, McNeil DW. A brief behavioral activation treatment for depression. A randomized pilot trial within an inpatient psychiatric hospital. Behav Modif. 2003 Sep;27(4):458-69. doi: 10.1177/0145445503255489. PMID 12971122
- [Background] Beck, AT, and Steer RA. Beck Hopelessness Manual. San Antonio, TX: The Psychological Corporation. 1988
- [Background] deJong Giervelde, J and Van Tilburg, TG. A six-item scale for overall emotional and social loneliness: Confirmative tests on a new survey data. Research on Aging, 28, 582-598, 2006.
- [Background] Mackenzie, CS, Knox, VJ, Gekoski, WL and Macaulay, HL. An adaption and extension of the Attitudes Toward Seeking Professional Psychological Help Scale. Journal of Applied Social Psychology, 34, 2410-2435, 2004.
- [Background] Ajzen, I. From intentions to actions: A theory of planned behavior. In J. Khul and J. Beckman (Eds). Action-control: From cognition to behavior (pp. 11-39) Heidelberg, Springer. 1985
- [Background] Cohen, J. Statistical power analysis for the behavioral sciences (2nd ed). Hillsdale, NJ, Lawrence Erlbaum Associates, 1988
- [Background] Luxton DD, Sirotin AP, Mishkind MC. Safety of telemental healthcare delivered to clinically unsupervised settings: a systematic review. Telemed J E Health. 2010 Jul-Aug;16(6):705-11. doi: 10.1089/tmj.2009.0179. PMID 20583951
- [Derived] Luxton DD, Pruitt LD, O'Brien K, Kramer G. An Evaluation of the Feasibility and Safety of a Home-Based Telemental Health Treatment for Posttraumatic Stress in the U.S. Military. Telemed J E Health. 2015 Nov;21(11):880-6. doi: 10.1089/tmj.2014.0235. Epub 2015 Jun 23. PMID 26103565

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In Home | In-Person
Started | 62 | 59
Completed | 40 | 42
Not Completed | 22 | 17
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Lost to Follow-up | 3 | 5
Not completed — randomized did not start treatment | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In Home | In-Person | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 59 | 121
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (12.4) | 35.6 (11.8) | 35.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 52 | 47 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 56 | 52 | 108
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 44 | 41 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 62 | 59 | 121

OUTCOME MEASURES:

1. Primary Outcome: Beck Hopelessness Scale (BHS)
Description: The BHS is a 20-item scale for measuring negative attitudes about the future. Each item is scored with a true/false response. Total scores range from 0-20 with higher scores indicating a greater degree of hopelessness.
Time Frame: Post treatment - Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 45 | 42
units on a scale | 4.888889 (4.642796) | 4.428571 (4.939353)
Statistical Analysis 1: Comparison: In Home vs In-Person; Test type: Non-Inferiority or Equivalence — One tailed test at .05a = .05 margin was set at standardized difference of .50; Regression, Beta = 0.40, 90% CI 2-sided [.12 to .68]

2. Secondary Outcome: Adverse Events
Description: Safety data will be collected on adverse events, psychiatric hospitalizations, suicides and non-fatal suicide-related behaviors, number of times the treatment collateral was utilized during treatment, treatment adherence, participant drop-out rate, and frequency of requests for patient or therapist technical support. Safety related data will be recorded after each treatment session on the Treatment Session Checklist.
Time Frame: Treatment Session Week 1
Population: AE data reported in adverse events section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
participants | 0 | 0

3. Secondary Outcome: Beck Depression Inventory -II (BDI-II)
Description: The BDI-II is the most commonly used self-report measure of clinical depression severity. It consists of 21 items that are rated on a 4-point scale which yield a range of scores from 0 - 63. The BDI-II has sound psychometric properties. The higher the score the worse the outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
units on a scale | 27.59678 (10.44652) | 29.71186 (11.33054)

4. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 2
Population: adverse event data reported in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
participants | 0 | 0

5. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 3
Population: adverse event data reported in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
participants | 62 | 59

6. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 4
Population: Adverse Event data recorded in Adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 48 | 44
participants | 0 | 0

7. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 5
Population: adverse events are reported in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 48 | 44
participants | 0 | 0

8. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 6
Population: adverse events are reported in the adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 48 | 44
participants | 0 | 0

9. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 7
Population: adverse events are reported in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 45 | 42
participants | 0 | 0

10. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: Treatment Session Week 8
Population: Adverse event data recorded in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 45 | 42
participants | 0 | 0

11. Secondary Outcome: Adverse Events
Description: as for outcome 2
Time Frame: 3 month follow up
Population: Adverse event data is recorded in adverse event section
Measure: Number; unit: participants
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 42 | 36
participants | 6 | 2

12. Secondary Outcome: Beck Depression Inventory -II (BDI-II)
Description: as for outcome 3
Time Frame: Midpoint- Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 47 | 44
units on a scale | 19.40425 (11.77444) | 20.20455 (13.09106)

13. Secondary Outcome: Beck Depression Inventory -II (BDI-II)
Description: as for outcome 3
Time Frame: Post Treatment- Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
units on a scale | 13.82222 (12.01947) | 11.7381 (12.07509)
Statistical Analysis 1: Comparison: In Home vs In-Person; Test type: Non-Inferiority or Equivalence — One tailed test at .05a = .05 margin was set at standardized difference of .50; Regression, Beta = .47, 90% CI 2-sided [.16 to .78]

14. Secondary Outcome: Beck Depression Inventory -II (BDI-II)
Description: as for outcome 3
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 42 | 36
units on a scale | 14.7619 (12.88752) | 15 (12.61065)

15. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 62 | 59
units on a scale | 9 (5.118273) | 10.37288 (6.133285)

16. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: as for outcome 1
Time Frame: Midpoint- Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 48 | 44
units on a scale | 7.041667 (5.63786) | 7.954545 (6.261564)

17. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: as for outcome 1
Time Frame: 3 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In Home | In-Person
Number analyzed (Participants) | 42 | 36
units on a scale | 5.214286 (5.101582) | 5.527778 (5.973686)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to final outcome assessment
Arm/Group | In Home | In-Person
Serious Adverse Events (participants affected / at risk) | 3/62 | 1/59
Other Adverse Events (participants affected / at risk) | 3/62 | 1/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Home (N=62) | In-Person (N=59)
exacerbation of asthma symptoms requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hospitalization for high fever and chills (Immune system disorders) | 1 (1) | 0 (0)
Severe chest pain (Cardiac disorders) | 0 (0) | 1 (1)
exacerbation of baseline suicidality (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Home (N=62) | In-Person (N=59)
broken nose (General disorders) | 1 (1) | 0 (0)
tore tendons in foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
syncopial episode (General disorders) | 1 (1) | 0 (0)
broken finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No